CLINICAL TRIAL: NCT01186497
Title: Relative Bioavailability of Rabeprazole Sodium Sprinkle Capsule Formulation Using Different Dosing Vehicles Following Single-dose Administration in Healthy Adult Subjects
Brief Title: A Relative Bioavailability Study of Rabeprazole Sodium Administered With Different Dosing Vehicles in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CR014821; RABGRD1004 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Healthy; Rabeprazole sodium; Rabeprazole sprinkle capsule granule formulation; Pharmacokinetics; Bioavailability; Safety; Adult

ARMS (5):
- Treatment sequence AEBDC (Experimental)
  Interventions: Drug: Rabeprazole sodium: Treatment E; Drug: Rabeprazole sodium: Treatment C; Drug: Rabeprazole sodium: Treatment D; Drug: Rabeprazole sodium: Treatment A; Drug: Rabeprazole sodium: Treatment B
- Treatment sequence BACED (Experimental)
  Interventions: Drug: Rabeprazole sodium: Treatment E; Drug: Rabeprazole sodium: Treatment C; Drug: Rabeprazole sodium: Treatment D; Drug: Rabeprazole sodium: Treatment A; Drug: Rabeprazole sodium: Treatment B
- Treatment sequence CBDAE (Experimental)
  Interventions: Drug: Rabeprazole sodium: Treatment E; Drug: Rabeprazole sodium: Treatment C; Drug: Rabeprazole sodium: Treatment D; Drug: Rabeprazole sodium: Treatment A; Drug: Rabeprazole sodium: Treatment B
- Treatment sequence DCEBA (Experimental)
  Interventions: Drug: Rabeprazole sodium: Treatment E; Drug: Rabeprazole sodium: Treatment C; Drug: Rabeprazole sodium: Treatment D; Drug: Rabeprazole sodium: Treatment A; Drug: Rabeprazole sodium: Treatment B
- Treatment sequence EDACB (Experimental)
  Interventions: Drug: Rabeprazole sodium: Treatment E; Drug: Rabeprazole sodium: Treatment C; Drug: Rabeprazole sodium: Treatment D; Drug: Rabeprazole sodium: Treatment A; Drug: Rabeprazole sodium: Treatment B

INTERVENTIONS:
Drug: Rabeprazole sodium: Treatment E — The contents of 2 rabeprazole sprinkle capsules equivalent to 10 mg rabeprazole sodium mixed with a tablet vehicle suspension (Treatment E) on Day 1.
Drug: Rabeprazole sodium: Treatment C — The contents of 2 rabeprazole sprinkle capsules equivalent to 10 mg rabeprazole sodium sprinkled on 1 tablespoon of applesauce (Treatment C) on Day 1.
Drug: Rabeprazole sodium: Treatment D — The contents of 2 rabeprazole sprinkle capsules containing 10 mg rabeprazole sodium mixed with 5 mL (1 teaspoon) of formula milk (Treatment D) on Day 1.
Drug: Rabeprazole sodium: Treatment A — The contents of 2 rabeprazole sprinkle capsules equivalent to 10 mg rabeprazole sodium mixed with a strawberry-flavored vehicle suspension (Treatment A) on Day 1.
Drug: Rabeprazole sodium: Treatment B — The contents of 2 rabeprazole sodium sprinkle capsules equivalent to 10 mg rabeprazole sodium sprinkled on 1 tablespoon of plain yogurt (Treatment B) on Day 1.

SUMMARY:
The purpose of the study is to investigate the bioavailability (rate and extent of absorption) of rabeprazole sodium when a sprinkle capsule granule formulation of rabeprazole sodium is mixed with different dosing vehicles (food, others) and is administered to healthy adult volunteers. Rabeprazole sodium is a drug used to treat patients with Gastro Esophageal Reflux Disease (GERD). GERD is a condition in which the esophagus (tube from throat to stomach) becomes irritated or inflamed because of acid backing up from the stomach.

DETAILED DESCRIPTION:
This is an open-label (volunteer and investigator will know the name of the assigned treatment) single center study to evaluate the bioavailability (rate and extent of absorption) and safety of different dosing vehicles used to administer a pediatric formulation of rabeprazole sodium to healthy adult volunteers. A dosing vehicle is a food or liquid that is mixed with rabeprazole sodium for oral (by mouth) administration. Approximately 35 healthy adult volunteers will be enrolled and randomized (assigned by chance) to 1 of 5 possible treatment sequences to receive each of the following single-dose treatments: 1) the contents of rabeprazole sprinkle capsules mixed in a strawberry-flavored vehicle suspension (Treatment A), 2) the contents of rabeprazole sprinkle capsules sprinkled on 1 tablespoon of plain yogurt (Treatment B), 3) the contents of rabeprazole sprinkle capsules sprinkled on 1 tablespoon of applesauce (Treatment C), 4) the contents of rabeprazole sprinkle capsules mixed with 5 mL (1 teaspoon) of formula milk (Treatment D), and 5) the contents of rabeprazole sprinkle capsules mixed in a tablet vehicle suspension (Treatment E). Each volunteer will receive 5 single-dose treatments during the study (1 single-dose treatment during each treatment period). A period of at least 7 days will separate each treatment period. During each treatment period, volunteers will be required to stay overnight at the study center for 12 hours before study drug administration up to approximately 24 hours after study drug administration to have study procedures performed and blood samples collected to measure the concentration of rabeprazole and its thioether metabolite (a substance produced when rabeprazole is absorbed in the body). Volunteers will fast (withhold from eating food) for at least 10 hours before study drug administration and up to at least 4 hours after study drug administration. On dosing days, volunteers will not receive a morning meal but will be allowed to drink non-carbonated water for up to 2 hours before study drug administration. After dosing, a standard lunch, snack, and dinner will be provided to volunteers. Each volunteer will participate in the study for approximately 55 days and be monitored for safety during the study by evaluating adverse events reported and results from clinical laboratory tests, 12-lead electrocardiograms (ECGs), vital sign measurements, and physical examinations. On Day 1 of each treatment period, volunteers will be administered the contents from 2 capsules equivalent to 10 mg of rabeprazole sodium mixed with a strawberry-flavored vehicle reconstituted with water or a vehicle tablet reconstituted with water (Treatments A and E, respectively) or 10 mg rabeprazole sodium sprinkled on 1 tablespoon of plain yogurt or applesauce (Treatments B and C, respectively), or 10 mg rabeprazole sodium mixed with 5 mL of formula milk (Treatment D).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers with a body mass index (ie, the relationship between a person's height and weight) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Have normal blood pressure between 90 and 140 mmHg systolic and <=90 mmHg diastolic
* Female volunteers must have a negative serum beta human chorionic gonadotropin (hCG) pregnancy test at screening and a negative urine pregnancy test on the day before each treatment period
* Female volunteers must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile, abstinent, or, if of childbearing potential and sexually active, be practicing an effective method of birth control before entry and throughout the study
* Male volunteers must agree to use an adequate contraception method as deemed appropriate by the investigator

Exclusion Criteria:

* Currently have, or have a history of clinically significant medical illness that the investigator considers should exclude the volunteer or that could interfere with the interpretation of the study results
* Have a history of drug or alcohol abuse within the past 1 year or a history of clinically significant allergies, especially known hypersensitivity or intolerance to milk products
* Have a history of smoking or use of nicotine-containing substances within the previous 2 months
* Have had major or traumatic surgery within 12 weeks before screening or preplanned surgery or procedures that would interfere with the conduct of the study
* known allergy to the study drug or any of the excipients of the formulation or known allergy to heparin or history of heparin-induced thrombocytopenia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Rabeprazole plasma concentrations | Day 1
Thioether metabolite plasma concentrations | Day 1

SECONDARY OUTCOMES:
The number of patients with adverse events as a measure of safety and tolerability | Approximately 55 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Thyssen A, Solanki B, Treem W. Randomized, open-label, single-dose, crossover, relative bioavailability study in healthy adults, comparing the pharmacokinetics of rabeprazole granules administered using soft food or infant formula as dosing vehicle versus suspension. Clin Ther. 2012 Jul;34(7):1636-45. doi: 10.1016/j.clinthera.2012.06.008. Epub 2012 Jun 29. PMID 22748970